CLINICAL TRIAL: NCT05811013
Title: Effects of Transcranial Static Magnetic Field Stimulation (tSMS) in Progressive Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Diego Centonze, Head of Neurology Unit, Neuromed IRCCS
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: tSMS-MS
Record Dates: First submitted 2023-03-16; First posted 2023-04-13 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Progressive Multiple Sclerosis
Keywords: Progressive Multiple Sclerosis; transcranial Static Magnetic Field Stimulation; disability progression; cortical hyperexcitability; cortical plasticity
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Intervention Model Description: We will conduct a randomized, sham-controlled, double-blind, within-subjects, cross-over study (allocation ratio 1:1) to test the ability of repeated sessions of tSMS to safely reduce disability progression in patients with PMS.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All patients, caregivers, and investigators assessing outcomes will be blind to the intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial static magnetic field stimulation (tSMS) (Experimental): Transcranial static magnetic field stimulation (tSMS) will be performed daily without any interruption during each session of 60 min. Each patient will be instructed to self-administer tSMS, two sessions per day (AM and PM, 6-10 hours apart), sequentially for 60 minutes each, for 6 +6 months.
  Interventions: Device: Transcranial static magnetic field stimulation (tSMS)
- Sham tSMS (Sham Comparator): Sham Transcranial static magnetic field stimulation (tSMS) Sham tSMS will be delivered with non-magnetic metal cylinders, with the same size, weight and appearance of the magnets (MAG45s; Neurek SL, Toledo, Spain). Real and sham magnets will be held with an ergonomic helmet (MAGmv1.0; Neurek SL, Toledo, Spain).
  Interventions: Device: Sham Transcranial static magnetic field stimulation (tSMS)

INTERVENTIONS:
Device: Transcranial static magnetic field stimulation (tSMS) — Patients will be randomly assigned to either real or sham tSMS. Real or sham tSMS will be performed daily without any interruption during each session of 60 min. Each patient will be instructed to self-administer tSMS, two sessions per day (AM and PM, 6-10 hours apart), sequentially for 60 minutes each, for 6 +6 months. Patients will choose whether to undergo stimulation at home or in the hospital on an outpatient setting. Real tSMS will be delivered with two cylindrical neodymium magnets (grade N45) of 45 mm diameter and 30 mm of thickness, with a weight of 360 g (MAG45r; Neurek SL, Toledo, Spain), applied with south polarity, each pointing toward the motor cortex. To discharge the weight of the helmet from the head during the sessions, patients will be instructed to rest the back of head and helmet on an inclined surface in a comfortable position. They will be also instructed to rest, minimizing movement, and not to watch audiovisuals during the stimulation sessions.
  Arms: Transcranial static magnetic field stimulation (tSMS)
Device: Sham Transcranial static magnetic field stimulation (tSMS) — Real or sham tSMS will be performed daily without any interruption during each session of 60 min. Each patient will be instructed to self-administer tSMS, two sessions per day (AM and PM, 6-10 hours apart), sequentially for 60 minutes each, for 6 +6 months. Sham tSMS will be delivered with non-magnetic metal cylinders, with the same size, weight and appearance of the magnets (MAG45s; Neurek SL, Toledo, Spain).
  Arms: Sham tSMS

SUMMARY:
In multiple sclerosis (MS) brains, inflammation induces specific abnormalities of synaptic transmission, collectively called inflammatory synaptopathy. Such synaptopathy consists in unbalanced glutamatergic and GABAergic transmission and in remarkable changes in synaptic plasticity, causing excitotoxic neurodegeneration and impairing the clinical compensation of the ongoing brain damage, thereby exacerbating the clinical manifestation of the disease. In progressive MS (PMS), synaptopathy is characterized by pathological potentatiation of glutamate-mediated synaptic up-scaling (Centonze et al., 2008; Rossi et al., 2013) and loss of long-term synaptic potentiation [LTP (Weiss et al., 2014)], both caused by proinflammatory molecules (released by microglia, astroglia, and infiltrating T and B lymphocytes) (Malenka et al., 2004; Di Filippo et al., 2017; Stampanoni Bassi et al., 2019). The combination of increased up-scaling and decreased LTP has a significant impact on the clinical manifestations of PMS, often presenting with signs and symptoms indicating length-dependent degeneration of neurons of the corticospinal tract. Altered LTP expression impairs brain ability to compensate ongoing neuronal loss (Stampanoni Bassi et al., 2020), and pathological TNF-mediated up-scaling may directly promote excitotoxic damage and neurodegeneration (Rossi et al., 2014). In addition, up-scaling and LTP are mutually exclusive at a given synapse through a mechanism of synaptic occlusion (i.e., pre-existing up-scaling saturates and prevents subsequent LTP expression), further promoting neurodegeneration by preventing the pro-survival effect of LTP, the induction of which activates intracellular anti-apoptotic pathways (Bartlett & Wang, 2013). It follows that a neuromodulation approach that can chronically (over several months) dampen up-scaling expression in the primary motor cortex (M1) of PMS patients could be beneficial by preventing excitotoxic neurodegenerative damage triggered by up-scaling itself (Centonze et al. 2008, Rossi et al. 2014), and also by promoting LTP induction and LTP-dependent functional compensation of deficits, thereby reducing the speed of the neurodegeneration process through increased LTP-dependent neuronal survival and preservation of dendritic spines (Ksiazek-Winiarek et al., 2015). Our study aims to test whether transcranial static magnetic field stimulation (tSMS) could represent such a therapeutic approach, as recently proposed in patients with amyotrophic lateral sclerosis (ALS) (Di Lazzaro et al, 2021). Forty (40) ambulatory patients with PMS, presenting with the ascending myelopathy phenotype of the disease, will be recruited at the MS Center of the Unit of Neurology of the IRCCS Neuromed in Pozzilli (IS). In this randomized, sham-controlled, double-blind, within-subjects, cross-over study (allocation ratio 1:1), we will test the ability of repeated sessions of tSMS applied bilaterally over the M1 to safely reduce disability progression in patients with PMS. Patients will be randomly assigned to either real or sham tSMS. Each patient will participate in two experimental phases (real or sham stimulation). Each patient will self-administer tSMS over right and left M1, two session per day, 60 minutes each. The order will be randomly established and counterbalanced across participants. Both investigators and participants will be blinded to stimulation parameters. In the "real stimulation" phase, tSMS will be applied for 120 minutes each day, at home, for 12 consecutive months. In the "sham stimulation" phase, sham tSMS will be delivered with non-magnetic metal cylinders, with the same size, weight and appearance of the magnets. Clinical evaluations, including the Multiple Sclerosis Functional Composite measure (MSFC) will be performed before, during and after each experimental phase ("real" and "sham"). In addition, blood levels of neurofilaments, excitability and plasticity of M1, and MRI measures of cortical thickness will be measured before, during and after each stimulation phase.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give written informed consent to the study
* Age range 18-65 years
* Diagnosis of primary of secondary progressive MS according to 2017 revised Macdonald's criteria (Thompson et al., 2017), presenting with signs of symptoms of progressive dysfunction of the corticospinal tract
* EDSS ≤ 6,5
* Ability to participate to the study protocol
* No or stable (at least six months) DMT or rehabilitative treatments before study entry, and willingness not to change these therapies (including cannabinoids, SSRI, baclofen) during the study.

Exclusion Criteria:

* Relapsing-remitting MS or progressive MS presenting with signs of symptoms other than those typical of the ascending myelopathy phenotype (i.e. progressive cerebellar or cognitive involvement)
* Female with positive pregnancy test at baseline or having active pregnancy plans
* Comorbidities for which synaptic plasticity may be altered (i.e., Parkinson's disease, Alzheimer's disease, stroke)
* Contraindications to TMS
* History or presence of any unstable medical condition such as malignancy or infection
* Use of medications with increased risk of seizures (i.e. Fampridine, 4-Aminopyridine)
* Concomitant use of drugs that may alter synaptic transmission and plasticity (L-dopa, antiepileptics)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-27 (Actual); Primary Completion 2025-05-27 (Estimated); Study Completion 2026-05-27 (Estimated)

PRIMARY OUTCOMES:
Functional assessment, that "change" is being assessed. | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  The primary aim the project is to evaluate the effect of tSMS in ambulatory patients with PMS with ascending myelopathy phenotype (from now on, simply called PMS) on clinical severity, assessed through the three components of the Multiple Sclerosis Functional Composite (MSFC).

SECONDARY OUTCOMES:
Neurological Assessment, that "change" is being assessed. | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Clinical severity will be assessed through the Expanded Disability Status Scale (EDSS).
Neuropsychological and psychometric evaluation | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Verbal episodic long-term memory will be evaluated with the Selective Reminding Test as LongTerm Storage (SeRT-LTS).
Neuropsychological and psychometric evaluation | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Verbal episodic long-term memory will be evaluated with the Consistent Long Term Retreival (SeRT-CLTR).
Neuropsychological and psychometric evaluation | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Verbal episodic long-term memory will be evaluated with the Delayed Recall (SeRT-DR).
Neuropsychological and psychometric evaluation | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Visuos patial episodic long-term memory will be evaluated with the Delayed Recall of Rey's Complex Figure (RCF- DR).
Neuropsychological and psychometric evaluation | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Executive functions and attention will be evaluated with Word List Generation (WLG).
Neuropsychological and psychometric evaluation | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Executive functions and attention will be evaluated with Symbol Digit Modalities Test (SDMT).
Neuropsychological and psychometric evaluation | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Executive functions and attention will be evaluated with Paced Auditory Serial Addition Test (PASAT).
Neuropsychological and psychometric evaluation | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Executive functions and attention will be evaluated with Stroop Test interference both in terms of errors (ST-E)
Neuropsychological and psychometric evaluation | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Executive functions and attention will be evaluated with response time (ST-RT)
Neuropsychological and psychometric evaluation | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Executive functions and attention will be evaluated with Brief Visuospatial Memory Test (BVMT)
Neuropsychological and psychometric evaluation | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Praxis ability will be evaluated with the Copy of Rey's Complex.
Neuropsychological and psychometric evaluation | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Anxiety will be assessed by State-Trait Anxiety Inventory form Y (STAI-Y)
Neuropsychological and psychometric evaluation | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Depression will be assessed with the Beck Depression Inventory-Second Edition (BDI-II).
Neurophysiological assessment | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Transcranial magnetic stimulation will be delivered with Magstim 2002 magnetic stimulators or with a Magstim Rapid2 stimulator (The Magstim Company, Whitland, Dyfed, UK). The stimulators will be connected to a figure-of-eight coil (external wing diameter 70 mm) placed tangentially over the scalp with the handle pointing back and away from the midline at about 45°, in the optimal position for eliciting motor evoked potentials (MEPs) in the first dorsal interosseous (FDI) muscle of the dominant hand. Electromyographic signals will be recorded with surface electrodes placed on the target muscle, sampled at 5 KHz with a CED 1401 A/D laboratory interface (Cambridge Electronic Design, Cambridge, UK), and amplified and filtered (bandpass 20 Hz to 2 kHz) with a Digitimer D360 amplifier (Digitimer Ltd, Welwyn Garden City, Hertfordshire, UK), then recorded by a computer with Signal software (Cambridge Electronic Design). Motor thresholds will be calculated at rest (RMT) as the lowest stimul
blood neurofilament light chain (NFL) levels | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Measures of NfL will be prospectively performed in the laboratory of Dr. Roberto Furlan (IRCCS San Raffaele, Milan). As a specific marker of neuroaxonal degeneration, increasing serum levels of NfL are seen in patients with a higher degree of disability independently of ongoing relapses (Bjornevik et al., 2020). Together with the medium and heavy subunits, NfL represents one of the scaffolding proteins of the neuronal cytoskeleton and is released in the extracellular space following axonal damage (Teunissen CE, Khalil M. 2012). The levels of serum sNfL, are a sensitive biomarker of ongoing neuroaxonal degeneration and represent a sensitive and clinically meaningful blood biomarker to monitor tissue damage and the effects of therapies in MS (Di Santo et al., 2017).
Magnetic Resonance Imaging (MRI) | BASELINE EVALUATION 1-30 DAYS BEFORE REAL OR SHAM tSMS T0; 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  Cortical thickness and T2 lesion load will be analyzed by using the 3T MR scanner (GE Signa HDxt, GE Healthcare, Milwaukee, Wisconsin). Will be used a 3D Spoiled Gradient Recalled (SPGR) T1-weighted sequence (178 contiguous sagittal slices, voxel size 1×1×1 mm, TR 7 ms, TE 2.856 ms, Inversion Time 450 ms) and a 3D FLAIR sequence (208 contiguous sagittal 1.6 mm slices, voxel size, 0.8 × 0.8 × 0.8 mm, TR 6000 ms, TE 139.45 ms; Inversion Time 1827 ms). White matter lesions will be segmented from FLAIR and T1 images by using the lesion growth algorithm as implemented in version 2.0.15 of the lesion segmentation tool (www.statistical-modelling.de/lst.html) for SPM12 (https://www.fl.ion.ucl.ac.uk/spm). Furthermore, the computational anatomy toolbox (CAT12, version 916, https://dbm.neuro.uni-jena.de/cat/) as implemented in SPM12 will be used to extract individual cortical thickness values from lesion-filled MR images. Finally, T2 lesion load will be computed from 3D T1 and 3d FLAIR images by
Patients' adherence to tSMS, potential side effects and adverse events | 6 MONTHS OF STIMULATION (SESSION 1, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 1, T12); 6 MONTHS OF STIMULATION (SESSION 2, T6); 1-30 DAYS AFTER THE END OF STIMULATION (SESSION 2, T12)
  The number of completed stimulation sessions will be recorded daily by each patient and/or the caregiver during the periods of self-administered tSMS treatment. Patients will fill a diary in which they will be instructed to record the following data:
  likert scale on sleep quality, presence of headache, treatment compliance. Potential side effects and adverse events will be reported by patients to the referring physician. If necessary, further clinical evaluations will be scheduled.
  At each timepoint, compliance will be assessed according to the following criteria:
  * "fully compliant" if he/she has performed at least 80% of the planned sessions of stimulation,
  * "moderately compliant" if he/she has performed between 50% and 80% of the treatment sessions,
  * "poor -compliant" if he/she has performed <50% of the treatment sessions. Caregivers will be instructed to monitor and favor treatment adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy

REFERENCES:
- [Background] Bartlett TE, Wang YT. The intersections of NMDAR-dependent synaptic plasticity and cell survival. Neuropharmacology. 2013 Nov;74:59-68. doi: 10.1016/j.neuropharm.2013.01.012. Epub 2013 Jan 25. PMID 23357336
- [Background] Bjornevik K, Munger KL, Cortese M, Barro C, Healy BC, Niebuhr DW, Scher AI, Kuhle J, Ascherio A. Serum Neurofilament Light Chain Levels in Patients With Presymptomatic Multiple Sclerosis. JAMA Neurol. 2020 Jan 1;77(1):58-64. doi: 10.1001/jamaneurol.2019.3238. PMID 31515562
- [Background] Bliss TV, Lomo T. Long-lasting potentiation of synaptic transmission in the dentate area of the anaesthetized rabbit following stimulation of the perforant path. J Physiol. 1973 Jul;232(2):331-56. doi: 10.1113/jphysiol.1973.sp010273. PMID 4727084
- [Background] Centonze D, Rossi S, Tortiglione A, Picconi B, Prosperetti C, De Chiara V, Bernardi G, Calabresi P. Synaptic plasticity during recovery from permanent occlusion of the middle cerebral artery. Neurobiol Dis. 2007 Jul;27(1):44-53. doi: 10.1016/j.nbd.2007.03.012. Epub 2007 Apr 5. PMID 17490888
- [Background] Di Filippo M, Mancini A, Bellingacci L, Gaetani L, Mazzocchetti P, Zelante T, La Barbera L, De Luca A, Tantucci M, Tozzi A, Durante V, Sciaccaluga M, Megaro A, Chiasserini D, Salvadori N, Lisetti V, Portaccio E, Costa C, Sarchielli P, Amato MP, Parnetti L, Viscomi MT, Romani L, Calabresi P. Interleukin-17 affects synaptic plasticity and cognition in an experimental model of multiple sclerosis. Cell Rep. 2021 Dec 7;37(10):110094. doi: 10.1016/j.celrep.2021.110094. PMID 34879272
- [Background] Di Lazzaro V, Profice P, Pilato F, Capone F, Ranieri F, Pasqualetti P, Colosimo C, Pravata E, Cianfoni A, Dileone M. Motor cortex plasticity predicts recovery in acute stroke. Cereb Cortex. 2010 Jul;20(7):1523-8. doi: 10.1093/cercor/bhp216. Epub 2009 Oct 5. PMID 19805417
- [Background] Di Lazzaro V, Musumeci G, Boscarino M, De Liso A, Motolese F, Di Pino G, Capone F, Ranieri F. Transcranial static magnetic field stimulation can modify disease progression in amyotrophic lateral sclerosis. Brain Stimul. 2021 Jan-Feb;14(1):51-54. doi: 10.1016/j.brs.2020.11.003. Epub 2020 Nov 10. No abstract available. PMID 33186779
- [Background] Disanto G, Barro C, Benkert P, Naegelin Y, Schadelin S, Giardiello A, Zecca C, Blennow K, Zetterberg H, Leppert D, Kappos L, Gobbi C, Kuhle J; Swiss Multiple Sclerosis Cohort Study Group. Serum Neurofilament light: A biomarker of neuronal damage in multiple sclerosis. Ann Neurol. 2017 Jun;81(6):857-870. doi: 10.1002/ana.24954. PMID 28512753
- [Background] Kos D, Kerckhofs E, Carrea I, Verza R, Ramos M, Jansa J. Evaluation of the Modified Fatigue Impact Scale in four different European countries. Mult Scler. 2005 Feb;11(1):76-80. doi: 10.1191/1352458505ms1117oa. PMID 15732270
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Ksiazek-Winiarek DJ, Szpakowski P, Glabinski A. Neural Plasticity in Multiple Sclerosis: The Functional and Molecular Background. Neural Plast. 2015;2015:307175. doi: 10.1155/2015/307175. Epub 2015 Jul 2. PMID 26229689
- [Background] Lu Y, Christian K, Lu B. BDNF: a key regulator for protein synthesis-dependent LTP and long-term memory? Neurobiol Learn Mem. 2008 Mar;89(3):312-23. doi: 10.1016/j.nlm.2007.08.018. Epub 2007 Oct 17. PMID 17942328
- [Background] Malenka RC, Bear MF. LTP and LTD: an embarrassment of riches. Neuron. 2004 Sep 30;44(1):5-21. doi: 10.1016/j.neuron.2004.09.012. PMID 15450156
- [Background] Mori F, Kusayanagi H, Nicoletti CG, Weiss S, Marciani MG, Centonze D. Cortical plasticity predicts recovery from relapse in multiple sclerosis. Mult Scler. 2014 Apr;20(4):451-7. doi: 10.1177/1352458513512541. Epub 2013 Nov 21. PMID 24263385
- [Background] Mori F, Rossi S, Piccinin S, Motta C, Mango D, Kusayanagi H, Bergami A, Studer V, Nicoletti CG, Buttari F, Barbieri F, Mercuri NB, Martino G, Furlan R, Nistico R, Centonze D. Synaptic plasticity and PDGF signaling defects underlie clinical progression in multiple sclerosis. J Neurosci. 2013 Dec 4;33(49):19112-9. doi: 10.1523/JNEUROSCI.2536-13.2013. PMID 24305808
- [Background] Rossi S, Studer V, Moscatelli A, Motta C, Coghe G, Fenu G, Caillier S, Buttari F, Mori F, Barbieri F, Castelli M, De Chiara V, Monteleone F, Mancino R, Bernardi G, Baranzini SE, Marrosu MG, Oksenberg JR, Centonze D. Opposite roles of NMDA receptors in relapsing and primary progressive multiple sclerosis. PLoS One. 2013 Jun 28;8(6):e67357. doi: 10.1371/journal.pone.0067357. Print 2013. PMID 23840674
- [Background] Rossi S, Motta C, Studer V, Macchiarulo G, Volpe E, Barbieri F, Ruocco G, Buttari F, Finardi A, Mancino R, Weiss S, Battistini L, Martino G, Furlan R, Drulovic J, Centonze D. Interleukin-1beta causes excitotoxic neurodegeneration and multiple sclerosis disease progression by activating the apoptotic protein p53. Mol Neurodegener. 2014 Dec 12;9:56. doi: 10.1186/1750-1326-9-56. PMID 25495224
- [Background] Rossi S, Motta C, Studer V, Barbieri F, Buttari F, Bergami A, Sancesario G, Bernardini S, De Angelis G, Martino G, Furlan R, Centonze D. Tumor necrosis factor is elevated in progressive multiple sclerosis and causes excitotoxic neurodegeneration. Mult Scler. 2014 Mar;20(3):304-12. doi: 10.1177/1352458513498128. Epub 2013 Jul 25. PMID 23886826
- [Background] Singer BH, Gamelli AE, Fuller CL, Temme SJ, Parent JM, Murphy GG. Compensatory network changes in the dentate gyrus restore long-term potentiation following ablation of neurogenesis in young-adult mice. Proc Natl Acad Sci U S A. 2011 Mar 29;108(13):5437-42. doi: 10.1073/pnas.1015425108. Epub 2011 Mar 14. PMID 21402918
- [Background] Stampanoni Bassi M, Iezzi E, Pavone L, Mandolesi G, Musella A, Gentile A, Gilio L, Centonze D, Buttari F. Modeling Resilience to Damage in Multiple Sclerosis: Plasticity Meets Connectivity. Int J Mol Sci. 2019 Dec 24;21(1):143. doi: 10.3390/ijms21010143. PMID 31878257
- [Background] Stampanoni Bassi M, Iezzi E, Mori F, Simonelli I, Gilio L, Buttari F, Sica F, De Paolis N, Mandolesi G, Musella A, De Vito F, Dolcetti E, Bruno A, Furlan R, Finardi A, Marfia GA, Centonze D, Rizzo FR. Interleukin-6 Disrupts Synaptic Plasticity and Impairs Tissue Damage Compensation in Multiple Sclerosis. Neurorehabil Neural Repair. 2019 Oct;33(10):825-835. doi: 10.1177/1545968319868713. Epub 2019 Aug 20. PMID 31431121
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Weiss S, Mori F, Rossi S, Centonze D. Disability in multiple sclerosis: when synaptic long-term potentiation fails. Neurosci Biobehav Rev. 2014 Jun;43:88-99. doi: 10.1016/j.neubiorev.2014.03.023. Epub 2014 Apr 12. PMID 24726576
- [Background] Yaka R, Biegon A, Grigoriadis N, Simeonidou C, Grigoriadis S, Alexandrovich AG, Matzner H, Schumann J, Trembovler V, Tsenter J, Shohami E. D-cycloserine improves functional recovery and reinstates long-term potentiation (LTP) in a mouse model of closed head injury. FASEB J. 2007 Jul;21(9):2033-41. doi: 10.1096/fj.06-7856com. Epub 2007 Mar 9. PMID 17351125
- [Background] Zepeda A, Aguilar-Arredondo A, Michel G, Ramos-Languren LE, Escobar ML, Arias C. Functional recovery of the dentate gyrus after a focal lesion is accompanied by structural reorganization in the adult rat. Brain Struct Funct. 2013 Mar;218(2):437-53. doi: 10.1007/s00429-012-0407-4. Epub 2012 Apr 6. PMID 22481229